CLINICAL TRIAL: NCT02631291
Title: A Randomized Pilot Study of Behavioral Self-monitoring to Promote Mental Health Among Spousally Bereaved Older Adults
Brief Title: Promoting Widowed Elders Lifestyle After Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sarah T. Stahl, PhD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PRO14110233
Record Dates: First submitted 2015-12-07; First posted 2015-12-16 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Mood Disorders; Depression; Anxiety; Grief; Bereavement; Health Behavior
MeSH Terms: conditions — Mood Disorders; Depression; Anxiety Disorders; Health Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lifestyle (Experimental): Behavioral self-monitoring of daily physical activity, dietary, and sleep behaviors, for 12 weeks, into an electronic tablet.
  Interventions: Behavioral: Behavioral self-monitoring
- Usual Care (No Intervention): Participants randomized to this condition will receive the written education provided to all participants.
- LIfestyle + coaching (Experimental): Behavioral self-monitoring of daily physical activity, dietary, and sleep behaviors, for 12 weeks, into an electronic tablet; and behavioral self-monitoring + motivational interviewing lifestyle coaching.
  Interventions: Behavioral: Behavioral self-monitoring + Motivational interviewing

INTERVENTIONS:
Behavioral: Behavioral self-monitoring — Behavioral self-monitoring will teach older adults to pay attention to their daily lifestyle practices and the conditions in which they occur. Behavioral self-monitoring is crucial for detecting change early, thereby preventing complications (mental illness symptom burden) that are associated with disruptions in healthy lifestyle practices. The steps of behavioral self-monitoring include: (1) selecting a goal, (2) paying attention to some aspect of behavior, and (3) recording some details of that behavior in a diary.
  Arms: Lifestyle
Behavioral: Behavioral self-monitoring + Motivational interviewing — Participants will receive the same Behavioral self-monitoring intervention; participants in this condition will interact with a 'lifestyle coach' about their recorded behaviors, weekly. The lifestyle coach will use motivational interviewing to enhance older adults' confidence and intrinsic motivation to engage in healthy lifestyle practices.
  Arms: LIfestyle + coaching

SUMMARY:
This study is for adults 60 years and older who are grieving the recent loss of a spouse or partner. Bereavement is one of the most distressing transitions faced by older adults and triggers dramatic changes to older adults' daily routine which puts them at-risk for a mood disorder. The purpose of this study is to promote bereaved elders' mental health by focusing on healthy lifestyle practices. Study treatment involves using a tablet to record their daily physical activity, diet, and sleep behaviors, for 12 weeks. The investigators follow-up with people for up to one year.

DETAILED DESCRIPTION:
Preventing mental health problems that develop following spousal bereavement is important because these conditions are highly prevalent and have lasting adverse consequences for the well-being of the bereaved survivor. The proposed research will evaluate the feasibility and acceptability of a healthy lifestyle intervention that uses a technology-based behavioral self-monitoring protocol to encourage engagement in physical activity, healthy eating, and good sleep practices following spousal bereavement. Data from 10 participants will be used for the development of a prevention intervention manual (Aim 1). A small pilot study will be conducted (Aim 2) in which 50 participants will be randomly assigned to 12 weeks of (1) behavioral self-monitoring using a smartphone (n=20), (2) behavioral self-monitoring using a smartphone + motivational interviewing-based lifestyle coaching (n=20), or (3) enhanced usual care (n=10). Blood samples will be collected to explore inflammatory cytokines as a potential mediator/moderator of mental health risk.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* experiencing the recent death (within 8 months) of a spouse or partner
* at-risk for developing mental health problems, based on high-risk markers defined as: subthreshold symptoms of depression (Hamilton Depression Rating Scale [HAM-D]101 of 9-14), anxiety (Generalized Anxiety Disorder Scale [GAD-7] ≥ 10, and/or complicated grief (Inventory of Complicated Grief [ICG] of 20-29), together with absence of current major depression, generalized anxiety, post-traumatic stress, or suicidiality; or high medical comorbidity (2 or more systems on the CIRS-G), low social support (Perceived Isolation Scale below zero), functional disability (limitation with at least 1 ADL/IADL),or

Exclusion Criteria:

* current DSM-V criteria for syndromal mood, psychosis, anxiety, eating disorder, or substance abuse dependence;
* dementia; 3MS<80;
* patients taking psychotropic medications to stabilize mental health problems including antidepressants and benzodiazepines;

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (Hamilton Rating Scale of Depression [HRSD]) | 12 months
  Symptom levels of depression (Hamilton Rating Scale of Depression [HRSD]),

SECONDARY OUTCOMES:
Anxiety symptoms (7-item Generalized Anxiety Disorder Scale [GAD-7]) | 12 months
  Symptom levels of anxiety (7-item Generalized Anxiety Disorder Scale [GAD-7])
Grief symptoms (Inventory of Complicated Grief [ICG]) | 12 months
  Symptom levels of complicated grief (Inventory of Complicated Grief [ICG])

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Stahl, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Sarah Stahl, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stahl ST, Croswell E, Patel K, Neagoe I, Minhaj S, Lopaczynski A, Lyew T. Long-term follow-up of clinical trial participants: Predictors of post-trial response in older subjects. Contemp Clin Trials. 2024 Aug;143:107579. doi: 10.1016/j.cct.2024.107579. Epub 2024 May 22. PMID 38789080